CLINICAL TRIAL: NCT02787174
Title: A Computer-Based ED Intervention to Improve Pediatric Asthma Medicine Adherence
Acronym: ED-AMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Aris Garro, Physician, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 629210; R21HD082621 (NIH)
Record Dates: First submitted 2016-05-19; First posted 2016-06-01 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: Asthma; Medication adherence; Intervention study
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Control (No Intervention): Participants will receive routine clinical treatment care.
- Intervention (Experimental): Participants will receive interactive tailored asthma medication adherence education on an iPad.
  Interventions: Other: Asthma Medication Adherence Education

INTERVENTIONS:
Other: Asthma Medication Adherence Education
  Arms: Intervention

SUMMARY:
Asthma is common in children and impacts their health. There are effective medications for improving asthma, but some families have difficulty using medicines on a regular basis. This study in the emergency department will improve medicine use for children 2-12 years-old with asthma by developing content for a customized, tablet-based electronic intervention. A clinical trial will then be used to compare asthma outcomes for this intervention with routine asthma care.

DETAILED DESCRIPTION:
The investigators have used focus groups to get ideas from parents of children with asthma to best design the intervention. This has helped us create the questions that are being used in the intervention, and make the computer program appealing and acceptable to parents of children with asthma.

The investigators will study the success of the intervention for children who receive it compared to children who obtain routine emergency department care. Participants who receive the intervention will complete a series of questions on a tablet computer. Questions will guide creation of individualized education and advice to improve medication use for each participant. The intervention will also allow for customized communication with each child's primary care provider. The investigators will include educational boosters at 2 and 4 weeks after the intervention delivered as chosen by the participant (email / text / RSS / mail). Children in the routine asthma care arm will not receive the intervention, and instead will receive routine discharge instructions by the emergency room doctors.

The investigators will compare the success of the intervention group to routine emergency department care by using a device (DOSER CT) that measures daily administered doses of medicine. Data from the DOSER CT will be collected monthly at home visits for three months. The investigators will also measure health care use and quality-of-life for each child using a survey at these home visits. The investigators believe that the intervention will improve doses of medicine given, reduce unnecessary health care use, and improve children's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis by physician or parent report
* Ages 2-12
* Prescribed an inhaled corticosteroid asthma controller medicine

Exclusion Criteria:

* Parent does not speak English
* Child is prescribed inhaled corticosteroid seasonally
* Patient is on a combination inhaled corticosteroid controller asthma med

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Asthma controller medication adherence | 12 weeks
  Percentage adherent days defined as at least half of prescribed doses taken as measured by Doser CT

SECONDARY OUTCOMES:
Unscheduled healthcare use (self-report survey and chart review) | 6 months
  Unscheduled healthcare use (Emergency Department visits, doctor visits, hospitalizations)
Quality-of-Life (QOL) | 6 months
  QOL measurement using Integrated Therapeutics Group Child Asthma Short Form (ITG-CASF)
Sustained Asthma controller medication adherence | 3 months
  Percentage adherent days defined as at least half of prescribed doses taken as measured by Doser CT

CONTACTS AND LOCATIONS:
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided